CLINICAL TRIAL: NCT01410006
Title: Neurofibromatosis Type 1 Patient Registry
Acronym: NPRI
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 10-1036
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Neurofibromatosis Type 1
Keywords: NF1; neurofibromatosis; NF
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibromatoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The Neurofibromatosis Type 1 (NF1) Patient Registry Initiative (NPRI) is a web-based registry that asks participants to fill out a 30-minute online questionnaire to collect information about the spectrum of medical and social problems experienced by children and adults with NF1. The information gained from your participation may one day help doctors develop personalized treatments for individuals living with NF1.

We are currently enrolling individuals with NF1 who either (1) HAVE previously been diagnosed with a brain tumor younger than 18 years or (2) HAVE NEVER had a brain tumor. Please note: there is no therapy associated with this study. Individuals may participate in the registry by going to https://nf1registry.wustl.edu/

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed by a healthcare provider with Neurofibromatosis Type 1

Exclusion Criteria:

* Individuals without a healthcare provider diagnosis of Neurofibromatosis Type 1

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is all individuals diagnosed with Neurofibromatosis Type 1.
Sampling Method: Non-Probability Sample
Enrollment: 2391 (Actual)
Dates: Start 2011-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Neurofibromatosis Type 1 | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly J Johnson, PhD, Study Director — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States